CLINICAL TRIAL: NCT04824326
Title: The Effects of Pythagorean Self-Awareness Intervention on Young Adolescents in Primary School-Α One Arm Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Aghia Sophia Children's Hospital of Athens (Other); Institute of Educational Policy (Unknown); Ministry of Education and Religions, Greece (Unknown)
Responsible Party: Principal Investigator, Orsalia Gerakini, Principal of 1st primary school,Neo Psychiko,Athens,Greece, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12413/09-11-2018
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Stress; Health Promotion; Adolescence
Keywords: holistic program; self-awareness; Pythagorean Self-Awareness Intervention; PSAI; stress; adolescence; school; bullying; healthy lifestyle; cognitive intervention
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pythagorean Self Awareness Intervention for Children and Adolescence(PSAI-CA) (Experimental): The intervention is based on the principles of the teaching of the ancient Greek philosopher Pythagoras. These principals set a basic framework for behavior on the basis of experiential learning and weekly evaluation of the implementation of 12 virtues. The technique is practiced twice a day(before night sleep and in the morning before getting up from bed) and evolves into five successive steps;1)reading of the 12 virtues and diaphragmatic breathing, 2)recall every event og the day,3)third person visualization and self-observation, 4)self-dialogue "What have I done wrong?", "What have I done right?", "What have I omitted that I ought to have done?" Endorsement or disapproval of actions according to the 12 virtues and the instructions for a healthy lifestyle, 5) next morning brief revision of the previous night's conclusions and setting of goals for the upcoming day.
  Interventions: Behavioral: PSAI-CA

INTERVENTIONS:
Behavioral: PSAI-CA — The intervention is based on the principles of the teaching of the ancient Greek philosopher Pythagoras. These principals set a basic framework for behavior on the basis of experiential learning and weekly evaluation of the implementation of 12 virtues. The technique is practiced twice a day(before night sleep and in the morning before getting up from bed) and evolves into five successive steps;1)reading of the 12 virtues and diaphragmatic breathing, 2)recall every event og the day,3)third person visualization and self-observation, 4)self-dialogue "What have I done wrong?", "What have I done right?", "What have I omitted that I ought to have done?" Endorsement or disapproval of actions according to the 12 virtues and the instructions for a healthy lifestyle, 5) next morning brief revision of the previous night's conclusions and setting of goals for the upcoming day.

SUMMARY:
In this one arm clinical trial, students of the 6th grade in a primary school participated in the PSAI for 8 weeks. Self-report questionnaires and hair cortisol concentrations were used for the evaluation of the aforementioned variables at baseline and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* attended the 6th Grade of primary education.

Exclusion Criteria:

* . absence of parental informed written consent
* diagnosis of mental health problemc.
* presence of any disease that could influence glucocorticoid levels
* pharmacological treatment that could influence cortisol levels
* practice of other stress management techniques

Ages: 12 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Stress reduction | Baseline-2months follow up
  Stress in Children (SiC) Questionnaire: This is a self-report psychometric instrument that consists of 21 items measuring physical, emotional and symptomatic aspects of stress in children. Each question is answered using a 4-point Likert-type scale (1 = never, 4 = very often). We expect reduction.

SECONDARY OUTCOMES:
Anxiety reduction | Baseline-2months follow up
  State-trait anxiety in children (STAIC): This is a "how-I-feel" questionnaire consisting of two forms of 20 items each which was designed as a research tool for the study of anxiety in children aged 9 to 12 years old. Half of the questions ask children how they feel at a particular moment in time responding to the state-anxiety scale, and the other half set of questions address how they usually feel responding to the trait-anxiety scale. Each item is answered using a 3-point Likert scale ranging from 3=very often to 1=rarely.We expect reduction.
Adherence to Mediterranean diet | Baseline-2months follow up
  KIDMED index: This is the Mediterranean diet quality index for children and adolescents which consists of 16 binary items(yes/no). Questions denoting a negative aspect regarding the MD were assigned a value of -1, and those with a positive one were assigned +1. We expect increase.
Amelioration of lifestyle | Baseline-2months follow up
  Healthy Lifestyle and Personal Control Questionnaire adapted for Children (HLPCQ): The HLPCQwas developed by the Postgraduate Course Stress Management and Health Promotion, School of Medicine, National and Kapodistrian University of Athens. Daily routine of the respondents was assessed with questions concerning (a) daily sleep, (b) breakfast, (c) lunch and (d) dinner and the regularity of components of their daily schedule Respondents were asked to give their answers ranging from 1 "never" to 4 "very often". Daily habits were assessed with a 4-point scale ranging from 1 "never" to 4 "always" for questions concerning eating habits, physical exercise, participation in sports, relations with relatives, support from friends. We expect increase.
Reduce bullying | Baseline-2months follow up
  Peer relations questionnaire for children (PRQ): The questionnaire was developed by Rigby and Slee (1993) and contains three subscales with 20 items. Bully subscale evaluates the tendency of a child to bully others and consists of 6 questions. The victim subscale evaluates the tendency to be victimized by others. The pro social subscale assessed the tendency to act in a pro social or cooperative manner. Four filler items are also included. Participants were asked to give their answers ranging from 1 "never" to 4 "very often". We expect reduction in victim-bully scales and increase in prosocial scale.
Investigation of hair cortisol concentrations | Baseline-3months followup
  Hair cortisol concentrations (HCC): The collection of hair tufts from each study participant took place at baseline and after three months (one month after completion of the intervention). From each participant, hair tuft was collected from the posterior vertexas close to the scalp as possible and stored in a paper envelope at room temperature, pending analysis. Collected hair segments were of one, up to multiple centimeters (cm) of length. Hair has a fairly predictable growth rate of about 1 cm/month. Therefore, the closest part of 1 cm to the scalp approaches the production of last month's cortisol. The second nearest 1 cm section approaches production during the month before, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Darviri, Study Director — National and Kapodistrian University of Athens, Greece
Locations (1):
- 4th primary school of Chalandri, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klinger DA, Freeman JG, Bilz L, Liiv K, Ramelow D, Sebok SS, Samdal O, Dur W, Rasmussen M. Cross-national trends in perceived school pressure by gender and age from 1994 to 2010. Eur J Public Health. 2015 Apr;25 Suppl 2:51-6. doi: 10.1093/eurpub/ckv027. PMID 25805788
- [Background] Lupien SJ, McEwen BS, Gunnar MR, Heim C. Effects of stress throughout the lifespan on the brain, behaviour and cognition. Nat Rev Neurosci. 2009 Jun;10(6):434-45. doi: 10.1038/nrn2639. Epub 2009 Apr 29. PMID 19401723
- [Background] Wigfield a, Lutz SL, Wagner AL. Early Adolescents' development across the Middle School Years: Implications for school Counselors. Professional School Counceling 2005;9(2):112-9. DOI:10.1177/2156759X0500900206
- [Background] Stults-Kolehmainen MA, Sinha R. The effects of stress on physical activity and exercise. Sports Med. 2014 Jan;44(1):81-121. doi: 10.1007/s40279-013-0090-5. PMID 24030837
- [Background] Simmons S, Limbers CA. Acculturative stress and emotional eating in Latino adolescents. Eat Weight Disord. 2019 Oct;24(5):905-914. doi: 10.1007/s40519-018-0602-2. Epub 2018 Oct 27. PMID 30367385
- [Background] Ouellet-Morin I, Wong CC, Danese A, Pariante CM, Papadopoulos AS, Mill J, Arseneault L. Increased serotonin transporter gene (SERT) DNA methylation is associated with bullying victimization and blunted cortisol response to stress in childhood: a longitudinal study of discordant monozygotic twins. Psychol Med. 2013 Sep;43(9):1813-23. doi: 10.1017/S0033291712002784. Epub 2012 Dec 10. PMID 23217646
- [Background] Takizawa R, Maughan B, Arseneault L. Adult health outcomes of childhood bullying victimization: evidence from a five-decade longitudinal British birth cohort. Am J Psychiatry. 2014 Jul;171(7):777-84. doi: 10.1176/appi.ajp.2014.13101401. PMID 24743774
- [Background] Kendall PC, Peterman JS. CBT for Adolescents With Anxiety: Mature Yet Still Developing. Am J Psychiatry. 2015 Jun;172(6):519-30. doi: 10.1176/appi.ajp.2015.14081061. PMID 26029805